CLINICAL TRIAL: NCT05422482
Title: An Open-Label, Phase 1 and Extension Study to Evaluate the Safety, Tolerability, PK and PD of Intracerebroventricular GC1123 in Patients with MPS Ⅱ Who Have Central Nervous System Involvement and Are Receiving Treatment with Intravenous Drug
Brief Title: A Study to Evaluate the Safety, Tolerability, PK and PD of Intracerebroventricular GC1123 in Patients with MPS Ⅱ
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC1123_MPS2_P0101
Record Dates: First submitted 2022-05-31; First posted 2022-06-16 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mucopolysaccharidosis II; Hunter Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GC1123 30mg (Experimental): 30 mg of IP will be administered every 28 days for all enrolled patients
  Interventions: Biological: GC1123

INTERVENTIONS:
Biological: GC1123 — ICV-administered Hunterase, Idursulfase-ß

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of intracerebroventricular GC1123 in patients with MPS Ⅱ who have central nervous system involvement and are receiving treatment with intravenous drug

DETAILED DESCRIPTION:
This study is designed as prospective, open-label, phase I and extension study. Safety, tolerability, pharmacokinetic, and pharmacodynamic properties of repeat-dose treatment of ICV-administered investigational product will be studied in patients undergoing standard treatments.

Patients will undergo cerebrospinal fluid (CSF) reservoir device implantation surgery on their scalps, and the reservoirs will be used to administer GC1123 to the cerebral ventricles monthly (every 28 days). The planned administering dose is 30 mg. After the 2nd dose on the 6th patient, Data and Safety Monitoring Boards (DSMB) will evaluate the safety and tolerability data of GC1123. The planned duration of the sutdy is total about 2 years (phase I and extension)

ELIGIBILITY:
Inclusion Criteria:

1. Patient who has been diagnosed with severe MPS Ⅱ (Hunter syndrome)
2. Patient, aged 1.5 years (18 months) to 18 years at the time of the screening
3. Patient who has received and tolerated a minimum of 12 weeks of treatment with weekly intravenous treatment, and who has received 80% of the total planned infusions within that time frame.
4. Patient who is capable of undergoing neurosurgery, which has been confirmed by neurosurgeons and anesthesiologist.
5. Patient eligible to execute patient evaluation activities during the clinical trial period, as assessed by the investigator
6. Patient whose parents or legal representative are willing to participate in this clinical trial and provide written informed consent form

Exclusion Criteria:

1. Patient who has been administered with intrathecal Idursulfase in the past
2. Patient with a history of bone marrow transplantation or cord blood transplant
3. Patient with a history of ventriculoperitoneal shunt or other intracranial surgeries
4. Patient with end-stage multiple organ dysfunction syndrome or other severe diseases
5. Patient who is exposed to malignant neoplasm
6. Patient who has received treatment with any investigational drug or device within 30 days prior to study entry
7. Patient who have experience of hypersensitivity or anaphylaxis to ingredients of the investigational product at the time of screening
8. Patient with a history of bronchotomy/tracheostomy, or patient with acute respiratory disease at the time of screening
9. Patient who is ineligible to participate in the clinical trial due to laboratory test results or other reasons, as determined by the investigator

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and frequency of serious adverse events (SAEs) | Every 28 days from Week 1 through study completion (about 110 weeks)
  Incidence and frequency of serious adverse events (SAEs) after administration of ICV-Hunterase (GC1123)
Frequency and characteristics (severity, outcome, etc.) of adverse events | Every 28 days from Week 1 through study completion (about 110 weeks)
  Frequency and characteristics (severity, outcome, etc.) of adverse events after administration of ICV-Hunterase (GC1123)
Presence of clinically significant abnormal echocardiography results | Week 1 to Phase I study completion (about 26 weeks)
  Presence of clinically significant abnormal echocardiography results after administration of ICV-Hunterase (GC1123); phase I only

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters - Cmax | Week 2 to Week 22
  Pharmacokinetic (PK) parameters of ICV-Hunterase (GC1123) in serum and CSF
Pharmacokinetic (PK) parameters - Tmax | Week 2 to Week 22
  Pharmacokinetic (PK) parameters of ICV-Hunterase (GC1123) in serum and CSF
Pharmacokinetic (PK) parameters - AUClast | Week 2 to Week 22
  Pharmacokinetic (PK) parameters of ICV-Hunterase (GC1123) in serum and CSF
Pharmacokinetic (PK) parameters - AUCinf | Week 2 to Week 22
  Pharmacokinetic (PK) parameters of ICV-Hunterase (GC1123) in serum and CSF
Pharmacokinetic (PK) parameters - t1/2 | Week 2 to Week 22
  Pharmacokinetic (PK) parameters of ICV-Hunterase (GC1123) in serum and CSF
Pharmacokinetic (PK) parameters - CL/F (or CL) | Week 2 to Week 22
  Pharmacokinetic (PK) parameters of ICV-Hunterase (GC1123) in serum and CSF
Pharmacokinetic (PK) parameters - Vd/F (or Vd) | Week 2 to Week 22
  Pharmacokinetic (PK) parameters of ICV-Hunterase (GC1123) in serum and CSF
Pharmacokinetic (PK) parameters - Bioavailability (F) | Week 2 to Week 22
  Pharmacokinetic (PK) parameters of ICV-Hunterase (GC1123) in serum and CSF
Pharmacodynamic (PD) parameters - Heparan Sulfate (HS) in CSF | Every 28 days from Week 1 through study completion (about 110 weeks)
  Pharmacodynamic (PD) parameters of ICV-Hunterase (GC1123)
Pharmacodynamic (PD) parameters - Heparan Sulfate (HS) in serum | Every 28 days from Week 1 through study completion (about 110 weeks)
  Pharmacodynamic (PD) parameters of ICV-Hunterase (GC1123)
Pharmacodynamic (PD) parameters - Urine Glycosaminoglycan (GAG) | Every 28 days from Week 1 through study completion (about 110 weeks)
  Pharmacodynamic (PD) parameters of ICV-Hunterase (GC1123)
Presence of anti-drug antibodies (ADAs) | Approximately every 6 months (Week 2 [baseline], Week 18, Week 26, Week 54, Week 82, Week 110)
  Presence of anti-drug antibodies (ADAs) in CSF and serum, and neutralizing antibodies of ICV-Hunterase (GC1123)

OTHER OUTCOMES:
Development Function assessed by Bayley Scales of Infant and Toddler Development-III and/or Kaufman Assessment Battery for Children-II (BSID-III/KABC-II) | Approximately every 6 months (Week 1 [baseline], Week 26, Week 54, Week 82, Week 110)
  All children will be tested for BSID-III, and children over the age of 3 will be also tested for KABC-II.
Adaptive Function assessed by Vineland Adaptive Behavior Scales 2nd Ed. (VABS-II) | Approximately every 6 months (Week 1 [baseline], Week 26, Week 54, Week 82, Week 110)
  Children under the age of 19 years will be tested for VABS-II.
Quality of Life (Survey) assessed by Infant and Toddler Quality of Life Questionnaire (ITQOL) and/or Childhood Health Questionnaire parent form (CHQ-PF50) | Approximately every 6 months (Week 1 [baseline], Week 26, Week 54, Week 82, Week 110)
  Children from the age of 2 months to 5 years will be tested for ITQOL, and children over the age of 5 will be tested for CHQ-PF50. The test performed during screening will be continued to be performed for each patient throughout the study period.
Liver and Spleen volume | Week 1 to phase I study completion (about 26 weeks)
  Liver and Spleen volume measured by MRI -phase I only

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Pusan National University Yangsan Hospital, Pusan
  - Seoul National University, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No